CLINICAL TRIAL: NCT05242354
Title: CD80, CD163 and CD206 Tissue Levels in Periodontal and Peri-implant Health and Disease
Brief Title: Macrophage Markers in Periodontal and Peri-implant Health and Disease
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Mustafa YILMAZ, Asst Prof, Biruni University
Other Study IDs: Peri-implant macrophage
Record Dates: First submitted 2022-01-28; First posted 2022-02-16 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Peri-Implantitis; Periodontitis
MeSH Terms: conditions — Peri-Implantitis; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Periodontal health: Periodontally healthy individuals (2017 Classification of Periodontal Diseases and Conditions) who are planned to receive crown lengthening / gingivectomy of tooth extraction involving at least one site with pocket depth ≤3mm, bleeding on probing -
- Peri-implant health: Periodontally healthy individuals (2017 Classification of Periodontal Diseases and Conditions) with at least one partially-exposed dental implant with no bone loss prior to the prosthetic rehabilitation
- Periodontitis: Generalized Stage III Grade C periodontitis patients (2017 Classification of Periodontal Diseases and Conditions) having at least one site with pocket depth ≥6mm, bleeding on probing +
- Peri-implantitis: Individuals with at least one implant site with radiographic bone loss, pocket depth ≥6mm and bleeding on probing +

SUMMARY:
Macrophage surface markers (CD80, CD163 and CD206) will be evaluated in periodontally healthy gingiva, healthy peri-implant mucosa, and periodontitis and peri-implantitis lesions.

DETAILED DESCRIPTION:
Soft tissue biopsies obtained from clinically healthy gingiva, healthy peri-implant mucosa, Stage III Grade C periodontitis lesions and peri-implantitis lesions will be evaluated.

Healthy peri-implant samples are obtained from submerged implants during exposure surgery. Healthy gingiva samples are obtained from individuals receiving crown lengthening, gingivectomy or tooth extraction as excess tissue during the corresponding treatment. Samples from peri-implantitis and periodontitis (pocket depth ≥6 mm, bleeding on probing+) are obtained during initial periodontal treatment / debridement procedure with a single stroke at the pocket wall.

The samples will be grinded and ultrasonicated. Western blotting will be used for determination of CD80, CD163 and CD206 in biopsy specimens. ImageJ will be used for intensity analysis of the bands.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with generalized Grade C Stage III periodontitis
* diagnosed with peri-implantitis
* periodontally healthy individuals with dental implants in the primary healing period
* periodontally healthy individuals who are in need of crown lengthening / gingivectomy or extraction

Exclusion Criteria:

* systemic disease
* smoking / former smokers
* regular medicine intake
* antibiotic or anti-inflammatory medicine intake in the last 3 months
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Otherwise healthy periodontitis, peri-implantitis patients or periodontally healthy individuals who applied to Biruni University Dentistry Faculty for treatment / regular oral examination
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to share the data with other researchers who demand it.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Periodontal Health | Peri-implant Health | Periodontitis | Peri-implantitis
Started | 10 | 8 | 9 | 9
Completed | 10 | 8 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Periodontal Health | Peri-implant Health | Periodontitis | Peri-implantitis | Total
Number analyzed (Participants) | 10 | 8 | 9 | 9 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 9 | 9 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11.7) | 44.4 (11.4) | 43 (18.8) | 48.7 (10.3) | 45.06 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 6 | 6 | 20
  Male | 5 | 5 | 3 | 3 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 10 | 8 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: CD80
Description: Tissue levels of CD80
  Western Blot assay analyzed using Image J software:
  Following scanning for optical densitometry, the gels were analyzed with Image J software by obtaining profile plots, drawing lines enclosing the interest area and measuring the peak area of interest with the wand tool. The calculated optical density values are presented as arbitrary density units.
Time Frame: Baseline
Measure: Median (95% Confidence Interval); unit: arbitrary density units
Units Other Than Participants: periodontal/peri-implant sites
Arm/Group | Periodontal Health | Peri-implant Health | Periodontitis | Peri-implantitis
Number analyzed (Participants) | 10 | 8 | 9 | 9
Number analyzed (periodontal/peri-implant sites) | 10 | 8 | 9 | 9
arbitrary density units | 7340.34 [3259.33 to 22949.08] | 10854.71 [6212.94 to 15352.85] | 6448.43 [4040.25 to 11881.73] | 9874.8 [5498.12 to 13903.64]

2. Primary Outcome: CD163
Description: Tissue levels of CD163
  Western Blot assay analyzed using Image J software:
  Following scanning for optical densitometry, the gels were analyzed with Image J software by obtaining profile plots, drawing lines enclosing the interest area and measuring the peak area of interest with the wand tool. The calculated optical density values are presented as arbitrary density units.
Time Frame: Baseline
Measure: Median (95% Confidence Interval); unit: arbitrary density units
Units Other Than Participants: periodontal/peri-implant sites
Arm/Group | Periodontal Health | Peri-implant Health | Periodontitis | Peri-implantitis
Number analyzed (Participants) | 10 | 8 | 9 | 9
Number analyzed (periodontal/peri-implant sites) | 10 | 8 | 9 | 9
arbitrary density units | 24092.85 [14131.26 to 39359.00] | 36419.24 [16424.64 to 40646.48] | 2167.97 [-2847.23 to 14877.20] | 6272.90 [1722.40 to 26614.33]

3. Primary Outcome: CD206
Description: Tissue levels of CD206
  Western Blot assay analyzed using Image J software (arbitrary density units):
  Following scanning for optical densitometry, the gels were analyzed with Image J software by obtaining profile plots, drawing lines enclosing the interest area and measuring the peak area of interest with the wand tool. The calculated optical density values are presented as arbitrary density units.
Time Frame: Baseline
Measure: Median (95% Confidence Interval); unit: arbitrary density units
Units Other Than Participants: periodontal/peri-implant sites
Arm/Group | Periodontal Health | Peri-implant Health | Periodontitis | Peri-implantitis
Number analyzed (Participants) | 10 | 8 | 9 | 9
Number analyzed (periodontal/peri-implant sites) | 10 | 8 | 9 | 9
arbitrary density units | 17648.07 [8965.15 to 25836.34] | 15063.13 [5505.74 to 37182.25] | 4049.07 [553.59 to 14523.94] | 16862.31 [8629.42 to 36697.95]

4. Primary Outcome: CD80/CD163 Ratio
Description: Tissue levels (Western Blot assay analyzed using Image J software) of CD80 divided by those of CD163
Time Frame: Baseline
Measure: Median (95% Confidence Interval); unit: ratio (no unit)
Units Other Than Participants: periodontal/peri-implant sites
Arm/Group | Periodontal Health | Peri-implant Health | Periodontitis | Peri-implantitis
Number analyzed (Participants) | 10 | 8 | 9 | 9
Number analyzed (periodontal/peri-implant sites) | 10 | 8 | 9 | 9
ratio (no unit) | 0.417 [0.139 to 0.902] | 0.413 [0.286 to 0.485] | 3.075 [1.338 to 5.135] | 0.801 [-0.792 to 8.762]

5. Primary Outcome: CD80/CD206 Ratio
Description: Tissue levels (Western Blot assay analyzed using Image J software) of CD80 divided by those of CD206
Time Frame: Baseline
Measure: Median (95% Confidence Interval); unit: ratio (no unit)
Units Other Than Participants: periodontal/peri-implant sites
Arm/Group | Periodontal Health | Peri-implant Health | Periodontitis | Peri-implantitis
Number analyzed (Participants) | 10 | 8 | 9 | 9
Number analyzed (periodontal/peri-implant sites) | 10 | 8 | 9 | 9
ratio (no unit) | 0.376 [-0.712 to 1.743] | 0.525 [0.283 to 1.232] | 1.366 [0.620 to 2.132] | 0.405 [-1.205 to 5.153]

6. Secondary Outcome: Probing Depth
Description: Probing depth of each site, where the tissue sample was harvested. The average probing depth of sites in each group are presented.
Time Frame: Baseline
Population: The probing depth of sites with periodontal health, periodontitis and peri-implantitis were recorded individually. Probing depth of the peri-implant health group was not measured, since the sites forming the peri-implant health group have no probable peri-implant sulcus/pocket.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal/peri-implant sites
Arm/Group | Periodontal Health | Periodontitis | Peri-implantitis
Number analyzed (Participants) | 10 | 9 | 9
Number analyzed (periodontal/peri-implant sites) | 10 | 9 | 9
mm | 1.5 (0.71) | 7.78 (0.83) | 7.78 (1.09)

ADVERSE EVENTS:
Time Frame: 6 months for periodontitis group one month for peri-implantitis group, peri-implant health group and periodontal health group
Arm/Group | Periodontal Health | Peri-implant Health | Periodontitis | Peri-implantitis
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05242354/Prot_SAP_000.pdf